CLINICAL TRIAL: NCT01309425
Title: A Single-Dose, Open-Label, Randomized, Four-Way Crossover Study to Assess the Dose-Proportionality of the Pharmacokinetics of Tapentadol, Given as Tamper-Resistant Tablets, in Healthy Japanese and Korean Male Subjects
Brief Title: A Study to Compare the Dose-proportionality of Tapentadol (CG5503) in Healthy Japanese and Korean Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CR017782; R331333PAI1064
Record Dates: First submitted 2011-03-03; First posted 2011-03-07 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2012-10

CONDITIONS: Healthy Volunteer
Keywords: tapentadol; NUCYNTA; CG5503; R331333; pharmacokinetics; healthy volunteer
MeSH Terms: interventions — Tapentadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 001 (Experimental): tapentadol (CG5503) ER 25-mg TRF 25mg TRF single oral dose
  Interventions: Drug: tapentadol (CG5503) ER 25-mg TRF
- 002 (Experimental): tapentadol (CG5503) ER 50-mg TRF 50mg TRF single oral dose
  Interventions: Drug: tapentadol (CG5503) ER 50-mg TRF
- 003 (Experimental): tapentadol (CG5503) ER 100-mg TRF 100mg TRF single oral dose
  Interventions: Drug: tapentadol (CG5503) ER 100-mg TRF
- 004 (Experimental): tapentadol (CG5503) ER two 100-mg TRF 200mg TRF single oral dose
  Interventions: Drug: tapentadol (CG5503) ER two 100-mg TRF

INTERVENTIONS:
Drug: tapentadol (CG5503) ER two 100-mg TRF — 200mg TRF single oral dose
  Arms: 004
Drug: tapentadol (CG5503) ER 50-mg TRF — 50mg TRF single oral dose
  Arms: 002
Drug: tapentadol (CG5503) ER 25-mg TRF — 25mg TRF single oral dose
  Arms: 001
Drug: tapentadol (CG5503) ER 100-mg TRF — 100mg TRF single oral dose
  Arms: 003

SUMMARY:
The purpose of this study is to evaluate the dose-proportionality of the pharmacokinetics of tapentadol (CG5503) in healthy Japanese and Korean adult male participants.

DETAILED DESCRIPTION:
This is a single-dose, open-label, single-center, randomized, four-way crossover study, ie, participants and investigator know the identity of the drug, which is assigned by chance, like flipping a coin, and participants may receive different interventions sequentially during the study. The study will consist of 4 treatment periods. A single dose of tapentadol (CG5503) will be administered orally with 240 mL of water under fasted conditions. All participants will receive 1 of the following 4 oral treatments in each period.

Treatment A: One 25-mg tablet (25 mg) of tapentadol (CG5503) Treatment B: One 50-mg tablet (50 mg) of tapentadol (CG5503) Treatment C: One 100-mg tablet (100 mg) of tapentadol (CG5503) Treatment D: Two 100-mg tablets (200 mg) of tapentadol (CG5503) Each period will be separated by 7 - 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese and Korean male volunteers, inclusive
* Body mass index (BMI) between 18.5 and 25 kg/m², inclusive, and a body weight of not less than 50 kg
* Japanese volunteers must have resided outside of Japan for no more than 5 years, and their parents and maternal and paternal grandparents are Japanese.
* Korean volunteers must have resided outside of Korea for no more than 5 years and their parents and maternal and paternal grandparents are Korean.

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease
* History of hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities
* History of significant pulmonary disease, including bronchospastic respiratory disease
* History of diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for paracetamol-acetaminophen, within 14 days before the first dose of the study drug is scheduled
* History of, or a reason to believe a participant has a history of drug or alcohol abuse within the past 5 years

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2011-02; Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile, as measured by Cmax, AUC, tmax, kel, t1/2 | Two days

SECONDARY OUTCOMES:
Number of participants with adverse events | Time of screening to end of treatment (up to 9.5 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.